CLINICAL TRIAL: NCT02891590
Title: Phase Ia Study of the Safety, Tolerability and PK of BTK Inhibitor DTRMWXHS-12 in Patients With B-Cell Lymphoma
Brief Title: Safety, Tolerability and PK of BTK Inhibitor DTRMWXHS-12 in Patients With B-Cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang DTRM Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTRM_DTRMWXHS-12_001
Record Dates: First submitted 2016-08-30; First posted 2016-09-07 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Chronic Lymphocytic Leukemia; B-cell Lymphomas
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — DTRMWXHS-12

ARMS (1):
- DTRMWXHS-12 (Experimental): DTRMWXHS-12 only: oral capsules (50 mg and 150 mg strengths), successive administration, dose escalation from 50mg to 100, 200, 400, 600, 800mg daily until MTD. During successive administration, orally once a day, 28 days as a cycle.
  Interventions: Drug: DTRMWXHS-12

INTERVENTIONS:
Drug: DTRMWXHS-12

SUMMARY:
The Primary Objective is to evaluate the safety and tolerability of multiple dose oral administration of DTRMWXHS-12 capsule in patients with B-cell lymphoma.

The Secondary Objective is to evaluate the pharmacokinetics of multiple dose oral administration of DTRMWXHS-12 capsule in patients with B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, gender is not limited. Patients are voluntary to sign the informed consent form.
* B-Cell Lymphoma based on WHO classified definition: including chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL); chronic lymphocytic leukemia with 17p-; mantle cell lymphoma (MCL); Waldenstrom's macroglobulinemia(WM); Diffuse large B-cell lymphoma (DLBL or DLBCL) etc.
* Measurable lesion: non-Hodgkin 's lymphoma requires at least a two-dimensional lesion diameter ≥ 2 cm, chronic lymphocytic leukemia ≥ 5000 leukemia cells / mm3, Waldenstrom's macroglobulinemia IgM ≥ 1000 mg / dL, bone marrow lymph plasma -like cells infiltration, Histopathologically diagnosed as Diffuse Large B- Cell Lymphoma.
* Investigator judges that the treatment is needed.
* Patients, who at least failed in lymphoma treatment once and without standard therapeutic options, can't satisfy the requirement or decline treatment or failed in autologous stem cell transplantation for Diffuse Large B- Cell Lymphoma.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 ~1
* Life expectancy greater than 4 months
* Ability to swallow capsules
* Hematologic functions satisfy: Neutrophils ≥1.5×109 / L ( according to the investigators' opinion , if they judge that the patients' neutrophil count lower than this threshold, which caused by chronic lymphocytic leukemia and bone marrow infiltration, those patients are eligible to be included. ), platelet(PLT) ≥75×109/L, HB≥80g/L
* Renal functions satisfy: Creatinine (Cr) ≤ 1.5 times of upper limit of normal persons; creatinine clearance rate≥50ml/min (estimated by Cockcroft-Gault formula or detected by nuclear medicine scan or 24 hours urine method)
* Liver functions satisfy: AST and ALT≤2.5 times of normal value, bilirubin ≤1.5 times of normal value
* Coagulation function: international normalized ratio (INR) and APTT ≤ 1.5 times of normal value;
* Throughout the course of the study and 90 days of treatment interruption, female of childbearing age and fertile males who must take one of the following effective contraception measures: abstinence, barrier-type dual contraceptive methods, IUDs, administration of hormonal contraception drug.
* Male subjects are prohibited sperm donation from the start to the end of treatment within 90 days.

Exclusion Criteria:

* Patients with brain metastasis
* Disease with changes of pathological tissue types (including large cell transformation)
* Patients who received allogeneic stem cell transplantation within 6 months, or with organized incompatibility reaction (GVHD), requires immunosuppressive therapy
* Patients who received steroid anti-tumor therapy within 7 days, or receive chemotherapy within 2 weeks, or receive monoclonal antibody therapy within 4 weeks, prior to first administration of DTRMWXHS-12 capsule.
* Patients received other BTK inhibitor therapy
* Patients had early received chemotherapy but their toxicity has not been cleared (according to NCI-CTCAE 4.03, unrecovered toxicity grade ≤1)
* Patients who received Chinese herbal anti-tumor therapy within 1 week before the start of study
* Patient with a history of other malignant within 2 years before enrollment, except (1) adequately treated in situ cervical cancer;(2) Local basal cell carcinoma or squamous cell carcinoma (3) Local malignant tumor which has been completely treated (by surgery or other means)
* Patients with uncontrolled systemic infection requiring intravenous anti-infection treatment
* Patients received major surgery in the past 4 weeks
* Patients with HIV infection, HBs-Ag positive
* According to New York Heart Association (NYHA) classification, patients with cardiovascular disease of grade ≥3
* Patients with history of Myocardial infarction, acute coronary syndrome (unstable angina), receiving coronary angioplasty and stent implantation within 6 months of study entry
* Patients applied something which may cause QT prolongation or accompany by torsades healer within 7 days prior to enrollment.
* Prolonged QTc interval (defined as a QTc> 450 ms) or other significant ECG abnormalities, including second degree atrioventricular block type Ⅱ, third degree atrioventricular block, or bradycardia (heart rate less than 50 beats / min),ECG QTc> 450 milliseconds, the ECG may be submitted to expert for centralized evaluation
* Subjects, the investigators think whose existing renal disease, neurological / psychiatric disorders, liver or endocrine disorders could affect their participating in the experiment
* Subjects with poor compliance
* Subjects are using CYP3A inhibitors (or inducer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Starting from date of first dose up to 30 days after last dose
  Confirm the safety and tolerability of multiple dose oral administration of DTRMWXHS-12 capsule

SECONDARY OUTCOMES:
Plasma concentrations of DTRMWXHS-12 | Days 1-28 (first treatment cycle)
  DTRMWXHS-12 Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, Ph.D., Study Director — Zhejiang DTRM Biopharma
Locations (1):
- Peking University Cancer Hospital, Beijing, China